CLINICAL TRIAL: NCT06351514
Title: An Open-Label, Single Arm Study of the Efficacy of Accelerated Intermittent Theta Burst Stimulation in Schizophrenia Patients With Persistent Negative Symptoms
Acronym: NOBLE-TMS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Mental Health, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023/00745
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia; Negative Type
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Accelerated iTBS — Patients will be assigned to receive iTBS over the left dorsolateral prefrontal cortex or Frontal Medea with 5 sessions a day, every weekday for 1 week and total of 25 sessions. Each iTBS session is approximately 10 minutes (depth corrected Resting Motor Threshold of 100%, 60 cycles of 10 bursts of three pulses at 50 Hz, repeated at 5 Hz; 2s on and 8s off; 1800 pulses per session; with a 50-minute interval between sessions. All TBS sessions will be performed by staff trained and credentialed in TMS according to Singapore College of Psychiatrists guidelines.

SUMMARY:
Schizophrenia patients commonly present with persistent negative symptoms which remain the main reason for dysfunction after recovery from an acute episode of psychotic symptoms. Negative symptoms in schizophrenia exact significant burden with no effective pharmacological or behavior treatment options thus far. Neuromodulatory modalities present a novel and alternative treatment approach and recent trials have shown preliminary evidence for the efficacy of intermittent Theta Burst Stimulation (iTBS) to treat negative symptoms in schizophrenia. In this study, we aim to examine the effectiveness of an accelerated iTBS treatment protocol as an augmentation treatment regime for patient in rehabilitation care with persistent negative symptoms.

We propose a pragmatic, open label and single arm clinical trial. Forty patients with diagnosis of schizophrenia, who had been stabilized from psychotic symptoms and currently suffering from dominant negative symptoms will be recruited and undergo accelerated iTBS treatment for 5 consecutive sessions each day for 5 working days. Participants will be followed up immediately, 1 month and 3 months after the end of treatment. Clinical assessment includes, BNSS, The Brief Negative Symptom Scale; SANS, Scale for the assessment of negative symptoms; SAPS, Scale for the assessment of positive symptoms; PANSS, Positive and Negative Symptoms Scale; MoCA, Montreal Cognitive Assessment scale; CDSS, Calgary Depression Scale for Schizophrenia: SDS, Sheehans' disability scale and EQ-5D. The primary endpoint of the trial is the change of negative symptoms as assessed by PANSS, negative symptoms subscale immediately after the treatment.

This study will determine whether accelerated iTBS is effective to be delivered as an augmentation therapy for patients with persistent negative symptoms. The optimal treatment system for this population can be immediately translated to clinical practice and benefit patients in need.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥21 and ≤65 years;
2. With primary diagnosis of schizophrenia or schizoaffective disorder;
3. Patients experienced prominent and persistent negative symptoms [Scale for the Assessment of Negative Symptoms (SANS) score ≥3 or Positive and Negative Symptoms Scale (PANSS)- negative subscale score ≥20] in past 6 months;
4. No clinically significant positive symptoms [PANSS positive subscale score <20];
5. No clinically significant depressive symptoms [Calgary Depression Scale for Schizophrenia (CDSS) score subscale <12];
6. Able to give consent.

Exclusion Criteria:

1. With current misuse of or dependence on illegal drugs or alcohol;
2. High Suicide risk;
3. History of epileptic seizures;
4. With severe brain trauma, injury or other neurological diseases;
5. Metal (implants) in the skull;
6. Pregnancy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change of Negative symptoms | Before treatment till Immediately post treatment.
  Assessed by PANSS, Negative symptoms subscale

SECONDARY OUTCOMES:
Trend of Negative symptoms | Before treatment till Immediately post treatment, 1 Month Post Treatment & 3 Month Post Treatment.
  Assessed by PANSS, Negative symptoms subscale

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Mental Health, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
Upon request, as approved by DSRB.